CLINICAL TRIAL: NCT00359840
Title: A Randomized, Dose - Finding Study of KRN321(Darbepoetin Alfa) for the Treatment of Anemia in Subjects With Solid Tumor
Brief Title: A Dose Finding Study of KRN321(Darbepoetin Alfa) for the Treatment of Anemia in Subjects With Solid Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KRN321-SC/05-A55
Record Dates: First submitted 2006-08-01; First posted 2006-08-03 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Anemia
Keywords: darbepoetin alfa; anemia; cancer patients; chemotherapy
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa

SUMMARY:
To assess the clinical effective dose of KRN321 administered with once triweekly schedule.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as solid tumor or malignant lymphoma
* patients receiving cyclic chemotherapy
* written informed consent
* hemoglobin concentration below 11 d/dL at enrollment
* life expectancy of more than 4 months

Exclusion Criteria:

* hemolysis, gastrointestinal bleeding, postoperative bleeding
* iron deficiency
* megaloblastic anemia
* received > 2 RBC transfusions within 4 weeks before randomization or any RBC transfusion within 2 weeks before randomization
* any primary hematological disorder that could cause anemia
* prior treatment with KRN321
* received erythropoetin therapy within 8 weeks before treatment

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To compare the effectiveness of KRN321(darbepoetin alfa) on the proportion of subjects achieving hemoglobin response

SECONDARY OUTCOMES:
To compare the proportion of subjects who receive red blood cell transfusions or show the hemoglobin level below 8 g/dL
To compare the proportion of subjects who receive red blood cell transfusions
To compare the effectiveness of KRN321 based on quality of life scores

CONTACTS AND LOCATIONS:
Overall Officials: Nagahiro Saijo, MD, Study Chair — National Cancer Center Hospital East
Locations (8):
- Japan (8):
  - Tokai region, Aichi
  - Shikoku region, Ehime
  - Kyusyu region, Fukuoka, Kumamoto
  - Hokkaido region, Hokkaido
  - Kinki region, Kyoto, Osaka, Nara
  - Tohoku region, Miyagi
  - Hokuriku region, Niigata, Ishikawa
  - Kanto region, Tochigi, Saitama, Tokyo, Kanagawa